CLINICAL TRIAL: NCT06740006
Title: Interest of Prefabricated Carbon Orthoses in the Therapeutic Arsenal of Children and Adolescents Affected by Central or Peripheral Neurological Pathologies: Retrospective Study on Gait Parameters and Prescription Criteria
Brief Title: Retrospective Study on the WalkOn AFO in Children or Teenagers With Neurological Pathologies
Status: Completed | Type: Observational
Sponsor: Otto Bock France SNC (Industry)
Responsible Party: Sponsor
Other Study IDs: BP-11-PT008
Record Dates: First submitted 2024-08-29; First posted 2024-12-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy (CP); Spastic Paraplegia; Spinal Cord Injuries (SCI); Spina Bifida; Neuropathy (Disorder)
MeSH Terms: conditions — Cerebral Palsy; Paraplegia; Spinal Cord Injuries; Spinal Dysraphism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to assess the interest of prefabricated carbon fiber ankle foot orthoses (AFO) in children and teenagers with central or peripheral neurological pathologies. The main question it aims to answer is:

Does prefabricated carbon AFO improve gait and provide user satisfaction? In current practice, all patients with gait impairments were fitted with this orthosis and had a 3D gait analysis with and without AFO. Biomecanical and follow-up data collected in current practice are analysed in this study in order to answer the question.

ELIGIBILITY:
Inclusion Criteria:

* Patient, child or adolescent, whose gait is affected by central or peripheral motor impairments
* Patient who has carried out a one-off trial of a WalkOn AFO (Ankle-Foot Orthosis) within the last 3 years prior to the beginning of the study (inclusion period)
* Patient whose quantified gait analysis with the WalkOn AFO and without orthosis is available in the medical file and whose date is within the inclusion period
* The investigator has verified that the patient and the parental authorities have received the information note concerning the study
* The investigator has verified that the person and the parental authorities do not object to the processing of data necessary for the study

Exclusion Criteria:

• Patients or holders of parental authority objecting to the processing of data within the framework of the study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children or tennagers whose gait is affected by central or peripheral motor impairments and who are followed in the rehabilitation center
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Stride length | After 1 hour with the device
  Biomechanical parameter: the distance between successive points of initial contact of the same foot (m)

SECONDARY OUTCOMES:
Walking speed | After 1 hour with the device
  Biomechanical parameter: the walking speed is the time one takes to walk a specified distance on level surfaces over a short distance (m/s).
Walking cadence | After 1 hour with the device
  Biomechanical parameter: the walking rate is equal to the walking speed divided by the stride lenth (steps/min).
Gait Profile Score | After 1 hour with the device
  Biomechanical parameter: the Gait Profile Score (GPS) is a clinical index that can be used to measure the overall deviation of gait data relative to normative data (°).
Gait Variable Score for the Hip | After 1 hour with the device
  Biomechanical parameter: the Gait Variable Score describes the joint specific measures of gait variability for the Hip (°).
Gait Variable Score for the Knee | After 1 hour with the device
  Biomechanicl parameter: the Gait Variable Score describes the joint specific measures of gait variability for the Knee (°).
Gait Variable Score for the Ankle | After 1 hour with the device
  Biomechanical parameter: the Gait Variable Score describes the joint specific measures of gait variability for the Ankle (°).
Walk ratio | After 1 hour with the device
  Biomechanical parameter: the walk ration represents the relationship between the amplitude and frequency of rhythmic leg movement during walking (m/step/min).
Antero-posterior Ground Force Reaction | Afer 1 hour with the device
  Biomechanical parameter: the antero-posterior Ground Force Reaction is the antero-posterior force exerted by the ground on a body in contact with it (N).
Time of Stance | After 1 hour with the device
  Biomechanical parameter: the time of stance is the time one spend with the foot on the floor (s)
Stance percentage | After 1 hour with the device
  Biomechanical parameter: the stance percentage is the percentage of time one spend with the foot on the floor during the gait cycle (%)
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | Between 3 to 18 months after the fitting with the device / Long-term follow-up visit
  Questionnaire: the QUEST measures the user satisfaction. It contains an evaluation part regarding the technology of the device on 8 items and one regarding services around the device on 4 items. It allows the patient to express himself on the criteria that are most important to him. An average satisfaction value can be calculated on a scale going from 1 to 5, with 1= "Not at all satisfied", 2="Not very satisfied", 3="more or less satisfied", 4="Quite satisfied" or 5="Very satisfied". The final QUEST score is the average obtained over all 12 items. Technology and services sub-scores can also be calculated.
  In this study, the french version ESAT (Evaluation des la Satisfaction envers une Aide Technique) is used.
  This questionnaire only concerns patients who purchase the orthosis, and was administered during a follow-up visit of the patient in the rehabilitation center.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Saint Pierre, Palavas-les-Flots, France

IPD SHARING:
Plan to Share IPD: No